CLINICAL TRIAL: NCT01158508
Title: Prophylactic Remote Ischemic Preconditioning for Cerebral Vasospasm Following Subarachnoid Hemorrhage
Brief Title: Remote Ischemic Preconditioning in Subarachnoid Hemorrhage
Acronym: RIPC-SAH
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-08-081-01
Record Dates: First submitted 2010-06-25; First posted 2010-07-08 (Estimated); Last update posted 2016-11-28 (Estimated); Status verified 2016-11

CONDITIONS: Subarachnoid Hemorrhage, Aneurysmal; Subarachnoid Hemorrhage; Cerebral Vasospasm; Intracranial Aneurysm
Keywords: cerebral aneurysm; cerebral vasospasm; subarachnoid hemorrhage; remote ischemic preconditioning
MeSH Terms: conditions — Subarachnoid Hemorrhage; Vasospasm, Intracranial; Intracranial Aneurysm

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Remote Ischemic Preconditioning (Experimental): Patients with aneurysmal subarachnoid hemorrhage, after aneurysm treatment, will be given prophylactic remote ischemic preconditioning by transient lower limb ischemia.
  Interventions: Procedure: Remote ischemic preconditioning

INTERVENTIONS:
Procedure: Remote ischemic preconditioning — Transient lower limb ischemia will be induced by inflation of a blood pressure cuff on the thigh. Four five minute cycles of ischemia will be performed, each followed by five minutes of reperfusion with the cuff down. This procedure will be performed in four rounds, typically on post-hemorrhage days 2, 3, 6 and 9.

SUMMARY:
Rupture of brain aneurysms is a common cause of death and disability, accounting for as many as 10% of stroke cases in the United States. While much of the resulting injury to the nervous system is caused by the initial bleeding from the aneurysm, many of these patients develop cerebral vasospasm, pathological constriction of the blood vessels supplying the brain, several days following hemorrhage. As many as a third of patients can suffer a resulting neurological deficit and stroke, presumably caused by the decreased blood flow to the brain (ischemia). This delayed brain injury accounts for a significant percentage of poor outcomes following aneurysm rupture. Studies have shown that remote ischemia to many organs can precondition other tissues (including the brain) to be more tolerant to decreases in blood flow. This "remote ischemic preconditioning" has the promise of protecting the brain from ischemic injury. Whereas in other forms of stroke the onset of ischemia cannot be predicted in the general population, following aneurysm rupture the investigators know which patients are likely to develop vasospasm and when. Therefore, ischemic preconditioning following aneurysm rupture may help prevent some of the ischemic injury caused by vasospasm. Remote ischemic preconditioning by transient limb ischemia (produced by inflation of a blood pressure cuff on the arm or leg) has been shown to minimize injury to other organs, most notably the heart. Remote ischemic preconditioning of the brain following aneurysm rupture has not yet been investigated.

DETAILED DESCRIPTION:
Phase I prospective clinical study to evaluate: the tolerance of clinical subjects with Subarachnoid Hemorrhage (SAH) to the maneuvers involved in the generation of Remote Ischemic Preconditioning (RIPC), the immediate and delayed hemodynamic effects of the RIPC in the cerebral vasculature, in terms of Transcranial Doppler (TCD) velocities, pulsatility index variations, Cerebral Blood Flow (CBF) measures, and cerebral arterial flow measurements using Magnetic Resonance Imaging with flow measurement capabilities (MRI NOVA). As a secondary goal, we will be valuating the impact of RIPC in the incidence of vasospasm, delayed neurological deficits, development of ischemic lesions in MRI and clinical outcome.

Patient Enrollment: Patients who are admitted to the University of California Los Angeles (UCLA) Ronald Reagan Medical Center with a diagnosis of aneurysmal subarachnoid hemorrhage will be considered for inclusion in this study. As is standard of care for this condition, following admission patients' aneurysms are generally treated by one of two methods, surgical clipping or endovascular coiling. Following this definitive treatment of the aneurysm, generally performed emergently in the first 24 to 48 hours following hemorrhage, patients will be consented and enrolled in the study. No patients with unprotected (untreated) aneurysms will be enrolled. Patients with a known history of lower limb vascular disease or lower limb vascular bypass surgery will be excluded.

Remote Ischemic Preconditioning (RIPC) Procedure: Following enrollment, patients will receive four rounds of lower limb remote ischemic preconditioning, starting at the earliest post-hemorrhage day possible following definitive treatment of their aneurysm. The remote ischemic preconditioning will typically take place on post-hemorrhage day 2, 3, 6 and 9. Each cycle of RIPC will consist of four 5-minute cycles of lower limb ischemia following by 5-minute periods of reperfusion. A large blood pressure cuff will be wrapped around the upper thigh of one leg. The cuff will be inflated to a pressure 20 mm Hg greater than the systolic arterial blood pressure measured by the patient's arterial line or upper limb blood pressure cuff. The adequate level of inflation will be confirmed by the absence of pulse in the ipsilateral pedal artery as detected by Doppler. The cuff will remain inflated for 5 minutes. The cuff will then be deflated and the limb will be allowed to re-perfuse for at least 5 minutes. After the cuff is deflated, the same procedure will then be repeated three times for a total of four cycles.

Evaluation of Tolerance to the RIPC Maneuvers: The patient will be continuously monitored for pain and discomfort during the RIPC session. If the patient pain is more than 6 in the traditional 1-10 scale or if the patient expresses their desire to stop the maneuver, the procedure will be stopped, and the data regarding number and duration of the maneuvers will be recorded. A down-escalation of the treatment will be proposed, by reducing the number of cuff inflations to 3 or 2, as tolerated.

Hemodynamic evaluation of the effect of RIPC Maneuvers: Transcranial Doppler (TCD) measurements will be performed during the RIPC session. TCD and Cerebral Blood Flow (CBF) measurements will be performed at 24 hours and 72 hours after treatment.

Cerebral arterial flow magnetic resonance imaging (MRI NOVA) will be measured the first day after treatment and 72 hours after treatment in patients suitable for transport to the MRI scan per Intensive Care Unit (ICU) clinical team criteria.

Clinical assessments of the patients will be performed daily and at discharge from the ICU

Treatment of subarachnoid hemorrhage (SAH) and Vasospasm: Aside from the RIPC procedures, all other treatment and monitoring of the patients will be as is standard of care for the treatment of patients with subarachnoid hemorrhage in our hospital. Patients will undergo neurological monitoring in the intensive care unit. Monitoring for cerebral vasospasm, including transcranial Doppler studies, angiograms, cerebral blood flow studies, Computed Tomography (CT) scans, Magnetic Resonance Imaging (MRI) scans and regular neurological examination will be performed as standard. Likewise, prophylaxis and treatment for vasospasm or any other complications of subarachnoid hemorrhage will be performed as usual, as is the standard of care. Apart from the rounds of RIPC, in no way will the monitoring and treatment of these patients differ from patients not enrolled in this study.

Data Collection: Patients' clinical data will be collected in a password-protected study computer database. General patient demographics, past medical history, history of present illness, Hunt & Hess grade, admission Glasgow coma score, modified Rankin score, size and location of aneurysm, dates of subarachnoid hemorrhage and aneurysm treatment, type of aneurysm treatment, transcranial Doppler study values, cerebral blood flow measurements, and results of clinical examinations will all be noted and recorded in the study database. Additionally, clinical imaging studies performed (including CT scans, MRI scans and cerebral angiograms) will be reviewed and their findings noted. Specifically, size and location of aneurysm, extent and location of subarachnoid hemorrhage, Fisher grade, and presence and size of ischemic brain lesions will be noted. Clinical complications and outcomes will be recorded, including occurrence of angiographic vasospasm and delayed neurological deficit and condition at discharge and follow-up (Glasgow outcome score and modified Rankin score). Any complications associated with the RIPC procedure will be noted and reported appropriately.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of recent aneurysmal subarachnoid hemorrhage.
* Definitive treatment of the aneurysm by surgical clipping or endovascular coiling has been completed.

Exclusion Criteria:

* Patients with unprotected (untreated) cerebral aneurysms.
* Patients with a known history of lower limb vascular disease, lower limb vascular bypass surgery and/or peripheral neuropathy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-04; Primary Completion 2014-01 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Occurrence of neurological events, or vasospasm | At days 3
Occurrence of neurological events, or vasospasm | At day 7
Occurrence of neurological events, or vasospasm | At day 15
Occurrence of neurological events, or vasospasm | At day 30

SECONDARY OUTCOMES:
Transcranial Doppler Measurements and metabolic assessment | At days 3
Transcranial Doppler Measurements and metabolic assessment | At day 7
Transcranial Doppler Measurements and metabolic assessment | At day 15

CONTACTS AND LOCATIONS:
Overall Officials: Nestor R Gonzalez, MD, Principal Investigator — University of California, Los Angeles David Geffen School of Medicine, Departments of Neurosurgery and Radiology
Locations (1):
- UCLA Ronald Reagan Medical Center, Los Angeles, California, United States

REFERENCES:
- [Result] Gonzalez NR, Connolly M, Dusick JR, Bhakta H, Vespa P. Phase I clinical trial for the feasibility and safety of remote ischemic conditioning for aneurysmal subarachnoid hemorrhage. Neurosurgery. 2014 Nov;75(5):590-8; discussion 598. doi: 10.1227/NEU.0000000000000514. PMID 25072112